CLINICAL TRIAL: NCT01400087
Title: Cap-attached Colonoscopy Versus Regular Colonoscopy for Trainees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Showa University (Other)
Responsible Party: Principal Investigator, Makoto Kutsukawa, Researcher, Showa University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: CAPSTUDY
Record Dates: First submitted 2011-07-21; First posted 2011-07-22 (Estimated); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Colonoscopy; Lower Gastrointestinal Tract
Keywords: colonoscopy; Lower Gastrointestinal Tract; Cecal intubation; Cap-attached colonoscopy; Trainee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cap-attached Colonoscopy (Active Comparator)
  Interventions: Device: Cap-attached Colonoscopy Versus Regular Colonoscopy
- Regular colonoscopy (Placebo Comparator)
  Interventions: Device: Cap-attached Colonoscopy Versus Regular Colonoscopy

INTERVENTIONS:
Device: Cap-attached Colonoscopy Versus Regular Colonoscopy — Trainees were divided into two group; Cap-attached Colonoscopy group or Regular Colonoscopy group. Trainees allocated to the former group undergo colonoscopy with cap for all cases, the latter without cap.

SUMMARY:
The aim of this prospective randomized controlled trial is to assess the efficacy of cap-attached colonoscopy to improve cecal intubation in comparison with regular colonoscopy for trainees.

DETAILED DESCRIPTION:
Colorectal cancer is one of the major malignancies in western countries and also in Japan. Therefore , the demand for total colonoscopy (TCS) has risen remarkably. However, failure to reach the cecum occurs in up to 10 % of cases.

A difficult colonoscopy procedure will often be associated with more complications, and require heavier sedation to alleviate patient's discomfort.

Auxiliary devices that could facilitate the examination would be needed. A cap is a simple device that can be attached to the tip of a colonoscope. The advantage of the cap in getting a good view might be helpful in cecal intubation by depressing the folds and also by keeping an appropriate distance between the colonoscope lens and colonic mucosa. We speculated that inexperienced colonoscopists would obtain greater benefit from cap-attached colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo colonoscopy examination

Exclusion Criteria:

* Known to have colonic stricture or obstructing tumor from the results of other investigations such as CT scan or barium enema
* Presence of acute surgical conditions such as severe colitis, megacolon, ischemic colitis and active gastrointestinal bleeding ・Patients who diagnosed as inflammatory bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
The success rate of cecal intubation | 24 hours

SECONDARY OUTCOMES:
The procedure time to achieve cecal intubation | 24 hours
Success rate in achieving terminal ileum intubation | 24 hours
The procedure time to achieve terminal ileum intubation | 24 hours
Complications related to the procedure | 24 hours
The dose of the intravenous drugs used | 24 hours
The polyp detection rate | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Shin-ei Kudo, Principal Investigator — Digestive Disease Center, Showa University Northern Yokohama Hospital
Locations (1):
- Digestive Disease Center, Showa University Northern Yokohama Hospital, Yokohama, Kanagawa, Japan

REFERENCES:
- [Background] Kondo S, Yamaji Y, Watabe H, Yamada A, Sugimoto T, Ohta M, Ogura K, Okamoto M, Yoshida H, Kawabe T, Omata M. A randomized controlled trial evaluating the usefulness of a transparent hood attached to the tip of the colonoscope. Am J Gastroenterol. 2007 Jan;102(1):75-81. doi: 10.1111/j.1572-0241.2006.00897.x. Epub 2006 Nov 13. PMID 17100978
- [Background] Lee YT, Lai LH, Hui AJ, Wong VW, Ching JY, Wong GL, Wu JC, Chan HL, Leung WK, Lau JY, Sung JJ, Chan FK. Efficacy of cap-assisted colonoscopy in comparison with regular colonoscopy: a randomized controlled trial. Am J Gastroenterol. 2009 Jan;104(1):41-6. doi: 10.1038/ajg.2008.56. PMID 19098847
- [Background] Harada Y, Hirasawa D, Fujita N, Noda Y, Kobayashi G, Ishida K, Yonechi M, Ito K, Suzuki T, Sugawara T, Horaguchi J, Takasawa O, Obana T, Oohira T, Onochi K, Kanno Y, Kuroha M, Iwai W. Impact of a transparent hood on the performance of total colonoscopy: a randomized controlled trial. Gastrointest Endosc. 2009 Mar;69(3 Pt 2):637-44. doi: 10.1016/j.gie.2008.08.029. PMID 19251004